CLINICAL TRIAL: NCT06848621
Title: A Single-blind, Randomized, Controlled Clinical Study of Flash Stimulation Therapy in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhang Baorong, Chief physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1021
Record Dates: First submitted 2025-02-04; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1:40Hz flash stimulation (Experimental): A one-week 40HZ flash stimulation therapy (JK-PMEG2700K light modulation glasses [light source]) using flash stimulation between 20:00 and 21:00.
  Interventions: Device: 40Hz light modulation glasses
- Group2:100Hz flash stimulation (Sham Comparator): A one-week 100HZ flash stimulation therapy (JK-PMEG2700K light modulation glasses [light source]) using flash stimulation between 20:00 and 21:00.
  Interventions: Device: 100Hz light modulation glasses

INTERVENTIONS:
Device: 40Hz light modulation glasses — A one-week flash stimulation therapy (JK-PMEG2700K light modulation glasses [light source]) using flash stimulation between 20:00 and 21:00.
  Arms: Group1:40Hz flash stimulation
Device: 100Hz light modulation glasses — A one-week flash stimulation therapy (JK-PMEG2700K light modulation glasses [light source]) using flash stimulation between 20:00 and 21:00.
  Arms: Group2:100Hz flash stimulation

SUMMARY:
The aim of this study was to evaluate the effect of flash stimulation therapy on the function of the cerebral glymphatic system and efficacy of improving symptoms in PD patients.

DETAILED DESCRIPTION:
Each subject will receive EEG recordings for two consecutive nights starting at 21:00. Participants will undergo baseline functional magnetic resonance imaging (fMRI). Subsequently, one week of flash stimulation therapy (JK-PMEG2700K light modulation glasses [light source]) was started, using flash stimulation between 20:00 and 21:00. After the 7-day flash stimulation treatment, a second round of clinical evaluation and fMRI will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. PD patients who meet the diagnostic criteria of the International Movement Disorders Association (MDS), between the ages of 50 and 70 years, the course of disease ≤5 years, and the Hoehn & Yahr stage ≤3;
2. Anti-PD drugs were taken regularly for at least one month before screening, and symptoms were stable;
3. The fixed bedtime in the past month is between 9:00 p.m. and 1:00 a.m., and the total sleep time is ≥6 hours;
4. Have the ability to understand and voluntarily sign informed consent;
5. Have good compliance and are willing to complete all follow-up required by this program.

Exclusion Criteria:

1. Secondary insomnia: including sleep disorders (restless leg syndrome, periodic limb movement disorder, sleep-related breathing disorders, etc.), physical diseases, mental disorders, psychoactive substance abuse;
2. suffering from photosensitive dermatitis, epilepsy and other diseases that are not suitable for flash stimulation;
3. Alcohol, coffee, or drug abusers in the past 6 months;
4. Mental illness: such as anxiety, depression, schizophrenia and post-traumatic stress disorder caused by insomnia;
5. Used drugs or health products that regulate sleep function or affect sleep within 14 days before enrollment or less than 5 drug half-lives;
6. Taking drugs that may impair cognitive ability, such as anticholinergic drugs, memory enhancing drugs, etc., within 7 days before enrollment;
7. the subject is unable to complete the test or follow-up;
8. suffering from other neurodegenerative diseases;
9. There are endoplants in the body that cannot be examined by MRI;
10. Inability to lie flat;
11. Other situations in which the researcher considers it inappropriate to participate in the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain glymphatic function | The first day after treatment
  The gBOLD-CSF coupling strength is improved in PD patients treated with 40Hz flash stimulation.

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale （MDS-UPDRS） | The first day after treatment
  MDS-UPDRS III score is decreased more than 3 points in PD patients treated with 40Hz flash stimulation.（The higher scores mean a worse outcome ）
Parkinson's disease sleep scale（PDSS） | The first day after treatment
  PDSS scale is decreased by more than 3 points in PD patients treated with 40Hz flash stimulation.（The higher scores mean a worse outcome ）

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
We will share the IPD when the article is published.